CLINICAL TRIAL: NCT03736265
Title: Clinical Study of Carvedilol for the Prevention of the Progression of Esophageal Varices in Hepatitis B Related Cirrhotic Patients With Anti-Viral Therapy
Brief Title: Carvedilol for Prevention of Esophageal Varices Progression
Acronym: Carvedilol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xiaojuan Ou, Director of liver research center, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017ZX10203202003
Record Dates: First submitted 2018-05-03; First posted 2018-11-09 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis, Liver; Portal Hypertension
Keywords: Portal Hypertension; Esophageal varices; Carvedilol
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol+ Nucleos(t)ide Analogues (Experimental): Based on nucleoside analogue (NUCs), carvedilol will added to the patients. Carvedilol is started at a dose of 6.25 mg once daily. After 1 week, this will increased to a dose of 12.5 mg once daily. Target dose of 12.5 mg once daily will be maintained if systolic blood pressure does not fall below 90 mm Hg and HR 50 beats per minute.
  Interventions: Drug: Carvedilol
- Nucleos(t)ide Analogues (No Intervention): Continuing take nucleoside analogue (NUCs) including lamivudine (LAM), adefovir dipivoxil (ADV), entecavir (ETV), telbivudine (TBV), tenofovir disoproxil fumarate (TDF) and tenofovir alafenamide (TAF).

INTERVENTIONS:
Drug: Carvedilol — Carvedilol is started at a dose of 6.25 mg once daily. After 1 week, this will increased to a dose of 12.5 mg once daily. Target dose of 12.5 mg once daily will be maintained if systolic blood pressure does not fall below 90 mm Hg and HR 50 beats per minute.
  Other Names: Nucleos(t)ide Analogues
  Arms: Carvedilol+ Nucleos(t)ide Analogues

SUMMARY:
Carvedilol has been shown to be more potent in decreasing portal hypertension to propranolol. But the efficacy of carvedilol to delay the growth of esophageal varices in chronic hepatitis B patients was unclear.

DETAILED DESCRIPTION:
It has been concluded 40%-70% of chronic hepatitis B patients can achieve fibrosis/ cirrhosis reversion after effective anti-viral therapy. But there is still some patients progress to decompensation. Esophageal varices are the main complication of cirrhotic patients. Propranolol are widely used to prevent variceal bleeding in patients with large esophageal varices. It has been shown the efficacy of propranolol in the preventing of the progression from small to large varices reported no effect. Recently, carvedilol has been shown to be more potent in decreasing portal hypertension to propranolol. But the efficacy of carvedilol to delay the growth of esophageal varices in chronic hepatitis B patients was unclear. The purpose of this study is to demonstrate the efficacy of carvedilol in the preventing of the progression from small to large varices in hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female;
* HBV-related liver cirrhotic patients with at least two years of antiviral therapy;
* The presence of small or medium esophageal varices without red color sign;
* HBV-DNA<1×10E3 IU/ml
* Signature of informed consent

Exclusion Criteria:

* Previous presence of decompensated cirrhosis including ascites, bleeding and HE (hepatic encephalopathy);
* Any contra-indications to beta-blockers including asthma, chronic obstructive pulmonary disease, allergic rhinitis, NYHA (New York Heart Association) class IV heart failure, atrioventricular block, sinus bradycardia (HR < 50 bpm), cardiogenic shock, hypotension (SBP < 90 mmHg), sick sinus syndrome, insulin dependent diabetes, peripheral vascular disease.
* Allergic to Carvedilol;
* Any malignancy that affects survival；
* Renal dysfunction；
* History of beta-blockers within last 3 months；
* History of surgery for portal hypertension；History of prior EVL (endoscopic variceal ligation) or sclerotherapy, history of surgery for portal hypertension including portosystemic shunts, disconnection and spleen resection and transjugular intrahepatic portosystemic shunt；
* Severe systemic diseases；
* Refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The progression Incidence of esophageal varices. | 2 years
  Progression of esophageal varices defines as follows:
  1. Varices developed from small(F1) to medium or large(F2/F3)
  2. Varices developed from medium(F2) to large(F3)
  3. Bleeding from esophageal varices.

SECONDARY OUTCOMES:
The incidence of liver cirrhosis decompensation | 2 years
  Cumulative rate of liver decompensation (including ascites,hepatic encephalopathy) after 2 year.
The incidence of hepatic cellular carcinoma, death or liver transplantation. | 2 years
  Cumulative rate of hepatic cellular carcinoma, death or liver transplantation after 2 year.
The progression rate of non-invasive scores (Child-Pugh、MELD、APRI、FIB-4 score). | 2 years
  The progression rate of Child-Pugh、MELD、APRI、FIB-4 score after 2 years.
The dynamic change of liver stiffness quantified by transient elastography. | 2 years
  The dynamic change of liver stiffness quantified by transient elastography after 2 years.
The dynamic change of hemodynamics parameter | 2 years
  The dynamic change of hemodynamics (HR and mean arterial pressure) after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Ou, Principal Investigator — Beijing Friendship Hospital
Locations (6):
- China (6):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang B, Zhou J, Wu X, Sun Y, Li L, Li P, Li M, Jiang W, Xu M, Feng B, Xu X, Cheng J, Xie W, Han T, Wang X, Li H, Piao H, Zhao X, Chen S, Meng T, Guan Q, Meng F, Kong Y, Ou X, Jia J, You H. Carvedilol Plus NUC for Patients With HBV-Compensated Cirrhosis Under Virological Suppression: A Randomized Open-Label Trial. Am J Gastroenterol. 2024 Apr 1;119(4):700-711. doi: 10.14309/ajg.0000000000002569. Epub 2023 Nov 6. PMID 37929952